CLINICAL TRIAL: NCT02320474
Title: Efficacy of Aflibercept (Eylea®) on Choroidal Neovascularization (Type 3)
Acronym: ATTRACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATTRACT
Record Dates: First submitted 2014-12-10; First posted 2014-12-19 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Type 3 Choroidal Neovascularization
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Experimental)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept

SUMMARY:
This is a one-year pilot, interventional, prospective, single arm, non-randomized, multicentric (3 centers) controlled study that aims to evaluate the response of type 3 choroidal neovascularization to treatment by Aflibercept following a classic protocol.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged more than 50 years
* Patients with type 3 choroidal neovascularization assessed on FA, ICG and OCT
* Exudation on SD-OCT scans defined by intraretinal cysts or subretinal fluid.
* Best Corrected Visual Acuity at inclusion between 24 and 78 letters (ETDRS)
* Media clarity, pupillary dilation and patient cooperation sufficient to allow fundus photographs of adequate quality

Exclusion Criteria:

* Any contraindications as reported in the labelling of Aflibercept (Eylea®): Ocular or periocular infection, Active intraocular inflammation or Hypersensitivity.
* Any previous history of intravitreal injections in the study eye for exudative AMD
* Any secondary chorioretinal anastomosis due to retinal scar or fibrosis
* Any history of vitrectomy
* Media opacities preventing accurate imaging of the retina (cataract)
* Any other retinal disorder possibly associated with type 3 CNV (epiretinal membrane, macular hole)
* Confirmed intraocular pressure ≥25 mmHg or non-stable glaucoma.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in Best Corrected Visual Acuity (BCVA) | 52 weeks
  Mean change from baseline in Best Corrected Visual Acuity (BCVA) as measured by ETDRS letter score at 4 meters

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas LEVEZIEL, MD, PhD, Principal Investigator — CHU Poitiers
Locations (2):
- France (2):
  - Poitiers University Hospital, Poitiers
  - Polyclinic of POITIERS, Poitiers